CLINICAL TRIAL: NCT00429039
Title: LLME Treated Cellular Immunotherapy Following T-cell Depleted Allogeneic Heamtopoietic Stem Cell Transplantation for Acceleration of Immune Reconstitution
Brief Title: A Study to Accelerate Immune System Recovery Following Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01.0082; 2000-66 (Other: CCRRC)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: L-leucyl-L-leucine methyl ester (LLME)

SUMMARY:
The purpose of this study is to determine if pre-treating donor lymphocytes with an investigational drug known as L-leucyl-L-leucine methyl ester (LLME, prior to donor lymphocyte infusion (DLI) will improve the recovery of the immune system following stem cell transplant.

DETAILED DESCRIPTION:
If you agree to participate in this research study you will be evaluated during the 4th-6th week after your transplant to determine the number of CD4 cells in your circulation and to determine that your body has eliminated all of the immune suppressing medicines used around the time of your transplant. This will be performed by studying the cells from two tubes of blood. Thereafter, blood cells will be obtained from your donor (the same donor as used for the transplant). These cells from the donor will be treated with LLME in the laboratory. The cells will then be washed to eliminate the LLME, counted, and the desired number will be administered to you by transfusion.

Four to six weeks later, you will have additional blood drawn (2-3 teaspoons) to determine the number of CD4 cells in your blood. If the number is below 100, you will be given another transfusion of LLME treated cells, but you will receive a larger number of cells. Above 100 CD4 cells, the risk of infections appears to decrease. This will be repeated every 8 weeks provided that you and your donor remain willing to continue until one of three things happens. The three things that would cause us to stop further DLI would be: (1) you develop a CD4 count of over 100, (2) you develop evidence of GVHD, or (3) we reach the maximum practical number of cells which your donor could provide.

Your donor will also be reevaluated by medical history, physical examination, and blood tests to ensure that he/she remains healthy and can undergo the cell donation procedure safely. He or she will donate the first doses of white cells by drawing a small amount of blood. Later donations, if necessary, will be collected in a manner that is very similar to how platelets are normally collected from volunteer donors by the blood bank. The manner in which the transfusions are given will be similar to that in which you have received red blood cell and platelet transfusions in the past.

ELIGIBILITY:
Inclusion Criteria:

* To be treated on this study, patients must have recently undergone a T-cell depleted allogeneic bone marrow or peripheral blood stem cell transplant from an HLA-matched sibling donor, an HLA matched unrelated donor, or an HLA partially matched (single antigen mismatched, two antigen mismatched, or haplodisparate) donor. Patients will be counseled and will sign informed consent for this study prior to their transplant. Our intention is to analyze the effectiveness of LLME treated DLI (Donor Lymphocyte Infusion) on an intent to treat basis. To proceed with this therapy after HSCT, patients must meet the other selection criteria below at the time of first DLI. Additionally, discussion prior to transplant helps present the patient (and donor) a picture of the proposed therapy in its entirety, rather than in piecemeal fashion. A patient or donor's unwillingness to participate in this study will in no way affect their eligibility for transplant therapy at our center.
* At the time of initial DLI therapy, patients must be between 28 and 42 days post allogeneic HSCT or between 28 and 42 days after the last dose of ATG if that agent was used after the transplant as part of their graft rejection prophylaxis. They must also meet the following criteria during the week prior to first infusion:
* Patients must have achieved primary engraftment with an absolute neutrophil count of at least 1000 per l for 3 consecutive days.
* Patients must have a CD4+ lymphocyte count of less than 200 per l. An absolute lymphocyte count of less than 200 per l will be taken as prime facie evidence that the CD4+ lymphocyte count meets this criteria.
* Patients may not exhibit overt hematologic manifestations of relapse or persistent disease. Evidence of recurrent/persistent disease based primarily on flow cytometry, cytogenetics, chimerism analysis, or other molecular studies does not by itself represent grounds for exclusion.
* Patients must be 16 years of age or older. There is no upper age limit for this study.
* Patients must not be pregnant.
* Patients must not have any documented graft-versus-host disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-09; Primary Completion 2007-10 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, M.D., Principal Investigator — Thomas Jefferson University, Department of Medical Oncology
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.KimmelCancerCenter.org